CLINICAL TRIAL: NCT05543759
Title: Simplified Combined Protocol for the Identification and Treatment of Acute Malnutrition in Venezuela
Brief Title: Simplified Treatment Protocol for Acute Malnutrition in Venezuela
Status: Terminated | Type: Observational
Why Stopped: The sponsoring organization UNICEF-Venezuela with administrative control over the study decided to terminate it.
Sponsor: UNICEF - Venezuela (Other)
Responsible Party: Sponsor
Other Study IDs: 291021
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Malnutrition in Childhood; Wasting; Child Malnutrition
Keywords: Severe acute malnutrition; Moderate acute malnutrition; Ready-to-use therapeutic food; Malnutrition treatment; Venezuela; Mid-upper arm circumference; Wasting
MeSH Terms: conditions — Cachexia; Child Nutrition Disorders; Severe Acute Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Children aged 6-59 months of both sexes from households established permanently in the catchment area of the selected health posts or health centers, meeting the SAM or MAM acute malnutrition case definitions described below with no medical complications and disability, and whose caregiver has granted consent to participate.
  Interventions: Dietary Supplement: Ready-To-Use Therapeutic Food (RUTF)

INTERVENTIONS:
Dietary Supplement: Ready-To-Use Therapeutic Food (RUTF) — * SAM [MUAC <115mm or WHZ <-3 or oedema (+/++)] = Two 92g sachets RUTF/day (Approx. 1000 kcal/day).
  * MAM [MUAC 115mm<125mm or WHZ <-2] = One 92g sachet RUTF/day (Approx. 500 kcal/day).

SUMMARY:
Global acute malnutrition (GAM) in children under five is defined by being too thin for a given height and/or having the Mid-upper arm circumference less than a given threshold. GAM includes moderate acute malnutrition (MAM) and severe acute malnutrition (SAM). This study has been designed to generate new evidence about the simplified combined protocol for the identification and treatment of GAM in Venezuela. The objective of the study is to document the safety and effectiveness of the Venezuelan simplified treatment protocol for GAM, which includes reduced frequency of follow-up visits, single product use and optimized daily RUTF dose. This prospective longitudinal study was conducted in 19 centers treating GAM in children aged 6-59 months diagnosed with uncomplicated GAM, defined as WHZ <-2 or MUAC <125mm or ++ bilateral edema. Children will be prospectively followed for a total of 6 months, including the treatment phase and the immediate post-discharge weeks until 6 months. The effectiveness of the treatment will be measured by the recovery rate, duration of the treatment and changes in anthropometry (weight, height and arm circumference). Other treatment effects will also be measured, including how many are admitted to the hospital, death and relapse rates from the nutritional program. An economic evaluation component will be incorporated. Total costs will be aggregated and presented as costs per child treated and per child recovered.

DETAILED DESCRIPTION:
The general objective of the study is to document the safety and effectiveness of Venezuelan simplified treatment protocol for Acute malnutrition of reduced frequency of follow-up visits, single product use and optimized daily RUTF dose.

This will be a prospective longitudinal study assessing the Venezuelan Simplified Combined Protocol among children with uncomplicated acute malnutrition according to the definition case study recently adopted by the Implementation Guidance: Prevention, Early Detection and Treatment of Wasting in Children 0-59 Months through National Health Systems in the Context of Coronavirus Disease, United Nations Children's Fund and World/Health Organization, for a single arm cohort included in treatment.

Children will be prospectively followed for a total of 6 months including the treatment phase and the immediate post-discharge weeks until 6 months.

An economic evaluation component will be incorporated. The economic valuation will be carried out based on quantitative data. Cost data will be collected from accounting records where available and through a series of interviews with key informants including health workers, civil society organizations, relevant staff from non-governmental organizations and United Nations agencies. Total costs will be aggregated and presented as cost per child treated and cost per child per child recovered.

The study will be implemented in 19 Community Health Centers purposively chosen based on their acute malnutrition prevalence and operational constraints. All of them will be proportionally distributed in three central states of Venezuela (Distrito Capital, Miranda, and La Guaira).

The protocol will be implemented by health professionals from each institution, duly previously trained in applying the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 6 and 23 months of age at inclusion.
* The mother must live in the study area from the time of inclusion.
* Mid-upper arm circumference (MUAC) <12.5 cm or WHZ <-2 or bilateral pitting edema.
* No serious medical complications.
* Positive appetite test.
* The consent of the mother or caregiver.

Exclusion Criteria:

* Congenital malformations that make anthropometric measurements impossible.
* Mother intends to leave the study area before six months.
* Presence of medical condition requiring referral for hospitalization.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible children are children aged 6-59 months of both sexes from households established permanently in the catchment area of the selected health posts or health centers, meeting the SAM or MAM acute malnutrition case definitions described above with no medical complications and disability, and whose caregiver has granted consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Recovery rate | Up to 4 months, from date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  This indicator is defined as the number children who recovered from wasting, MAM and SAM according to national program criteria (WHZ>-2 and MUAC>=125mm and absence of bilateral edema for two consecutive visits, within 16 weeks of enrollment in the program) divided by the total number of treatment results recorded.
Weight gain | Up to 4 months, from date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average weight change per month
MUAC gain | Up to 4 months, from date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average change in MUAC per month
Duration of the treatment | Up to 4 months, from date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Defined as the average number of weeks spent on treatment (enrollment and discharge) in children 6-59 months of age at enrollment, according to health registers
Prevalence of relapse after discharge from the treatment | at six months after the admission
  This indicator is defined as the proportion of children with WHZ-score <-2 or MUAC <125 mm or bilateral edema six months after the admission
Number of RUTF delivered per child | Up to 4 months, from date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average number of RUTF delivered per child (SAM/MAM)
Cost per child | Up to 4 months, from date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average number of dollars that cost to recovery a child

SECONDARY OUTCOMES:
Longitudinal prevalence of wasting | Up to 6 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  This indicator is defined for each child as the number of visits during which nutritional wasting is observed divided by the total number of monthly visits made.
Prevalence of child stunting | Up to 6 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Proportion of children with Height-for-age Z-score (LAZ)<-2 (according to the 2006 World Health Organization reference) at the end of the study
Prevalence of child morbidity | Up to 6 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Defined by the number of days with symptoms of acute respiratory infections, fever, diarrhea (three or more loose or liquid stools per day) and malaria divided by the total number of days observed/reported in the recall period
Prevalence of readmission | Up to 6 months, at 24 weeks after the admission
  Prevalence of children readmitted to the treatment within six months after after the admission

CONTACTS AND LOCATIONS:
Overall Officials: Zulay Gonzalez, MSc, Principal Investigator — UNICEF - Venezuela
Locations (1):
- Distrito Capital, La Guaira, Miranda, Caracas, Distrito Federal, Venezuela

IPD SHARING:
Plan to Share IPD: No